CLINICAL TRIAL: NCT03430635
Title: What is the Prognostic Value of ¹¹C-choline PET/CT in Patients Undergoing Hepatectomy for Hepatocellular Carcinoma?
Brief Title: Role of Choline PET/CT in Predicting Survival in Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Assistant Professor of Surgery, Humanitas Clinical and Research Center
Other Study IDs: CholinePETforHCC
Record Dates: First submitted 2018-01-20; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hepatectomy — Surgery of the liver: removal of a given part of the liver affected by hepatocellular carcinoma
  Other Names: Hepatic resection; liver resection.

SUMMARY:
¹¹C-choline positron emission tomography/computed tomography (PET/CT) has been used in patients with some types of solid cancers, but few data are available in patients undergoing hepatectomy for hepatocellular carcinoma (HCC). The aim of this study was to analyze the prognostic value of metabolic imaging data by using ¹¹C-choline PET/CT in patients with HCC before hepatectomy.

DETAILED DESCRIPTION:
Our prospectively maintained liver unit database was queried for patients with HCC preoperatively staged with ¹¹C-choline PET/CT. This metabolic imaging modality was performed in addition to standard abdominal CT or magnetic resonance imaging. Several PET/CT parameters were recorded and analyzed. Univariate and multivariate analyses were performed to identify whether those PET/CT parameters could be predictors of overall survival (OS) and disease-free survival (DFS) of HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with HCC candidate to surgical resection preoperatively staged with ¹¹C-choline PET/CT

Exclusion Criteria:

* R2 resection;
* Intraoperative use of RFA/MWI
* Postoperative death (90-days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by HCC candidate to surgical resection that were preoperatively staged with ¹¹C-choline PET/CT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Identification of PET/CT parameters that can be predictors of survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first assessed up to 72 months
  Identification of specific PET/CT parameters that can be used as independent predictors of overall and/or disease-free survival

REFERENCES:
- [Background] Lanza E, Donadon M, Felisaz P, Mimmo A, Chiti A, Torzilli G, Balzarini L, Lopci E. Refining the management of patients with hepatocellular carcinoma integrating 11C-choline PET/CT scan into the multidisciplinary team discussion. Nucl Med Commun. 2017 Oct;38(10):826-836. doi: 10.1097/MNM.0000000000000719. PMID 28723716
- [Background] Lopci E, Torzilli G, Poretti D, de Neto LJ, Donadon M, Rimassa L, Lanza E, Sabongi JG, Ceriani R, Personeni N, Palmisano A, Pedicini V, Comito T, Scorsetti M, Chiti A. Diagnostic accuracy of (1)(1)C-choline PET/CT in comparison with CT and/or MRI in patients with hepatocellular carcinoma. Eur J Nucl Med Mol Imaging. 2015 Aug;42(9):1399-407. doi: 10.1007/s00259-015-3079-5. Epub 2015 May 12. PMID 25962590